CLINICAL TRIAL: NCT04326439
Title: CHOA-AML: A Pilot Study for Newly Diagnosed Pediatric Patients With Acute Myeloid Leukemia (AML)
Brief Title: AflacLL1901 (CHOA-AML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to unforeseen circumstances, the study team was limited in enrolling patients on this trial; thus, it was terminated.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Himalee Sabnis, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00111627
Record Dates: First submitted 2020-03-13; First posted 2020-03-30 (Actual); Results first posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia; AML, Childhood
Keywords: acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; Asparaginase; asparaginase erwinia chrysanthemi recombinant; Etoposide; Gemtuzumab; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Bone Marrow Transplantation; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aflac-AML Regimen for Low Risk AML Patients (Experimental): Participants in this arm will receive the standard Aflac-AML Regimen with the following chemotherapy:
  * Induction-1: patients on Induction-I will receive gemtuzumab + ADE therapy based on genotyping. Lasts a total of 28 days.
  * Induction II - MA
  * Intensification I - AE
  * Intensification II - HD ARAC/LASP
  Patients with low risk status who had low risk markers and were MRD positive at the end of Induction I and continue to be MRD positive after Induction II will come off protocol.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Erwinase; Drug: Etoposide; Drug: Gemtuzumab ozogamicin
- Aflac-AML Regimen for High Risk AML Patients (Experimental): Participants in this arm will receive standard Aflac-AML Regimen with the following chemotherapy:
  * Induction-1: patients will receive gemtuzumab in addition to ADE therapy based on genotyping. Induction I lasts a total of 28 days.
  * Induction 1 for FLT3-ITD patients - ADE (10+3+5) with GO with Sorafenib
  * Induction II - MA
  * Induction II for FLT3-ITD patients - MA with Sorafenib
  * Intensification I - AE
  * Intensification I for FLT3-ITD patients - AE with sorafenib
  * Intensification II - HD ARAC/LASP
  * Intensification II for FLT3-ITD patients - HD ARAC/LASP with sorafenib
  * Hematopoietic stem cell transplantation (HSCT)
  If a patient is classified as High risk after Induction I, they may proceed to best allogenic donor SCT following Induction II. These patients may receive a third course of chemotherapy prior to HSCT. In cases where HSCT is not an option, patients can receive 4 cycles of chemotherapy. Only patients with FLT3-ITD mutation will receive sorafenib.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Erwinase; Drug: Etoposide; Drug: Gemtuzumab ozogamicin; Procedure: Stem cell transplantation (SCT); Drug: Sorafenib

INTERVENTIONS:
Drug: Cytarabine — 100 mg/m²/dose every 12 hours IV Days 1-10
  Other Names: cytosine arabinoside, ARA-C
Drug: Daunorubicin — 50 mg/m²/dose IV Days 1, 3, 5
  Other Names: Rubidomycin
Drug: Erwinase — 25,000 International Units/m²/dose IM Days 2, 9
  Other Names: Erwinaze, Erwinia L-Asparaginase, Erwinia Chrysanthemi L-asparaginase, Crisantaspase
Drug: Etoposide — 150 mg/m²/dose IV Days 1-5
  Other Names: VePesid, VP-16
Drug: Gemtuzumab ozogamicin — Administered as a single 3 mg/m2 dose of GO to be given between days 6-10 during Induction I for patients with CC genotype, in addition to ADE therapy.
  Other Names: Mylotarg®, CDP-771, CMA-676, hP67.6-calicheamicin
Procedure: Stem cell transplantation (SCT) — Transplantation of multipotent hematopoietic stem cells from bone marrow
  Other Names: Hematopoietic stem cell transplantation (HSCT), Bone Marrow Transplant (BMT)
  Arms: Aflac-AML Regimen for High Risk AML Patients
Drug: Sorafenib — 200 mg/m2/dose daily, rounded to accommodate tablet size. The maximum dose will be 400 mg. Days 7 through 34.
  Other Names: BAY 43-9006 Tosylate, BAY 54-9085 Nexavar
  Arms: Aflac-AML Regimen for High Risk AML Patients

SUMMARY:
The investigators propose to study an Aflac-AML chemotherapy backbone prospectively to validate its use in all pediatric AML and to further evaluate the cardiotoxicity with this approach for low risk AML.

DETAILED DESCRIPTION:
Advances in risk stratification and therapy, have improved the event-free survival (EFS) and overall survival (OS) for pediatric acute myeloid leukemia (AML) to approximately 50% and 65% respectively, with current treatment strategies. Patients with good response to induction and/or those who lack high-risk cytogenetic and molecular features [classified as low-risk AML (LR-AML)] have even better outcomes with EFS and OS approaching 70% and 85% respectively; however, treatment-related toxicities remain a major concern. Anthracycline-based therapeutic regimens expose patients to the risk of anthracycline-induced cardiotoxicity. Therefore, strategies that reduce cardiac toxicities using tailored approaches while maintaining and/or improving outcomes are needed for all patients with AML. The Children's Oncology Group (COG) regimens AAML1031 and AAML0531 utilized an anthracycline-intensive backbone for LR-AML with cumulative anthracycline doxorubicin-equivalent doses of up to 492mg/m2. However, high-risk patients treated with chemotherapy alone received an intensified induction chemotherapy (using mitoxantrone-cytarabine) but with overall reduced doses of anthracycline-equivalent (342mg/m2). The investigators piloted an institutional practice to treat all LR-AML patients with four cycle regimen (Aflac-AML) with the goal of reducing cumulative anthracycline exposure, thereby reducing the risk of cardiotoxicity, while providing three high-dose cytarabine courses. In this pilot institutional experience with this approach, they were able to maintain excellent outcomes for this low-risk group with 3-year event-free survival (EFS) and OS of 70.0% ± 0.1% and 85.5% ± 0.08% respectively, from end of course 1. Recent evolution in cytogenetic classification has further delineated risk groups in AML. Gemtuzumab ozogamicin (GO), an antibody-drug conjugate was shown to reduce relapse risk in patients with CC genotype with de-novo AML on COG study AAML0531. The investigators propose to study an Aflac-AML chemotherapy backbone prospectively to validate its use in all pediatric AML and to further evaluate the cardiotoxicity with this approach for low risk AML.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be less than 21 years of age at the time of study enrollment
* Diagnosis: Patients must be newly diagnosed with AML
* Patients with previously untreated primary AML who meet the customary criteria for AML with ≥ 20% bone marrow blasts as set out in the 2016 WHO Myeloid Neoplasm Classification are eligible.
* Attempts to obtain bone marrow either by aspirate or biopsy must be made unless clinically prohibitive. In cases where it is clinically prohibitive, peripheral blood with an excess of 20% blasts and in which adequate flow cytometric and cytogenetics/FISH testing is feasible can be substituted for the marrow exam at diagnosis.
* Patients with <20% bone marrow blasts are eligible if they have:

  * A karyotypic abnormality characteristic of de novo AML (t(8;21)(q22;q22), inv(16)(p13q22) or t(16;16)(p13;q22) or 11q23 abnormalities,
  * the unequivocal presence of megakaryoblasts, or
  * Biopsy proven isolated myeloid sarcoma (myeloblastoma; chloroma, including leukemia cutis)
* Performance Level: Patients with acceptable organ function and any performance status are eligible for enrollment

Exclusion Criteria:

* Patients with any of the following constitutional conditions are not eligible:

  * Fanconi anemia
  * Shwachman syndrome
  * Any other known bone marrow failure syndrome
  * Patients with constitutional trisomy 21 or with constitutional mosaicism of trisomy 21 Note: Enrollment may occur, pending results of clinically indicated studies to exclude these conditions.
* Other Excluded Conditions:

  * Any concurrent malignancy
  * Juvenile myelomonocytic leukemia (JMML)
  * Philadelphia chromosome positive AML
  * Biphenotypic or bilineal acute leukemia
  * Acute promyelocytic leukemia (APL)
  * Acute myeloid leukemia arising from myelodysplasia
  * Therapy-related myeloid neoplasms

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himalee Sabnis, MD, Principal Investigator — Emory University
Locations (1):
- Egleston Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabnis HS, Minson KA, Monroe C, Allen K, Metts JL, Cooper TM, Woods WG, Castellino SM, Keller FG. A strategy to reduce cumulative anthracycline exposure in low-risk pediatric acute myeloid leukemia while maintaining favorable outcomes. Leuk Res. 2020 Sep;96:106421. doi: 10.1016/j.leukres.2020.106421. Epub 2020 Jul 12. PMID 32683126

RESULTS

PARTICIPANT FLOW:
Groups:
- Aflac-AML Low Risk Patients: Patients were classified as low risk following Induction I. All were MRD negative without low or high risk genetic and prognostic factors.
  * Induction I: AraC/Daunorubicin/Etoposide (10+3+5) +/- GO based on CC genotype
  * Induction II: Mitoxantrone/AraC
  * Intensification I: AraC/Etoposide
  * Intensification II: HD AraC/Asparaginase
- Aflac-AML High Risk Patients: Patients were classified as high risk following Induction I. All were MRD negative with high risk genetic and prognostic factors.
  Induction I: AraC/Daunorubicin/Etoposide (10+3+5) +/- GO based on CC genotype^ Induction II: Mitoxantrone/AraC^ Intensification:* AraC/Etoposide^ OR HD AraC/Asparaginase^ Allogenic HSCT
  * ^If has FLT3-ITD mutation, Sorafenib is added
  * * Depending on timing patients may proceed to HSCT following Induction II or receive Intensification. If HSCT is not an option, patients can receive 4 cycles of chemotherapy
Period: Overall Study
Arm/Group | Aflac-AML Low Risk Patients | Aflac-AML High Risk Patients
Started | 5 | 3
Completed | 3 | 0
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Proceeded to HSCT after Induction 2 | 0 | 2
Not completed — Relapse after Induction 2 | 0 | 1
Not completed — Refractory CNS Leukemia after 6 doses IT cytarabine | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflac-AML Low Risk Patients | Aflac-AML High Risk Patients | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.8 (0.8) | 4.1 (4.4) | 2.7 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) in Low Risk Patients and High Risk Patients
Description: Event-free survival defined as the time from on study to death, failure to achieve remission or relapse in newly diagnosed patients with pediatric acute myeloid leukemia in the Low risk stratification group and High risk stratification group
Time Frame: Up to 2 years post-intervention
Measure: Median (Full Range); unit: years
Arm/Group | Aflac-AML Low Risk Patients | Aflac-AML High Risk Patients
Number analyzed (Participants) | 5 | 3
years | 1.20 [0.16 to NA] — Insufficient number of participants with events; maximum observation was censored at last follow-up. | 0.76 [0.23 to NA] — Insufficient number of participants with events; maximum observation was censored at last follow-up.

2. Secondary Outcome: Overall Survival (OS)
Description: Time from study entry and from end of first course of therapy for newly diagnosed patients with pediatric acute myeloid leukemia
Time Frame: Up to 2 years post-intervention
Measure: Median (Full Range); unit: years
Arm/Group | Aflac-AML Low Risk Patients | Aflac-AML High Risk Patients
Number analyzed (Participants) | 5 | 3
years | 1.97 [0.36 to NA] — Insufficient number of participants with events; maximum observation was censored at last follow-up | 1.98 [0.21 to NA] — Insufficient number of participants with events; maximum observation was censored at last follow-up

3. Secondary Outcome: Minimal Residual Disease (MRD) Negative Status
Description: Number of patients that are in remission (MRD negative) after course 1 in participants receiving GO and those that did not receive GO.
Time Frame: Post-induction I, an average of 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Induction I With GO: Patients with CC genotype received Induction 1 AraC/Daunorubicin/Etoposide (10+3+5) with Gemtuzumab ozogamicin (GO)
- Induction I Without GO: Patients without CC genotype received Induction 1 AraC/Daunorubicin/Etoposide (10+3+5)
Arm/Group | Induction I With GO | Induction I Without GO
Number analyzed (Participants) | 5 | 3
Participants | 5 | 3

4. Secondary Outcome: Disease-free Survival (DFS) for Patients Who Are MRD Negative
Description: Disease-free survival for patients who are MRD negative but lack high or low risk molecular and cytogenetic features, defined as time from end of first course of therapy to death or relapse
Time Frame: Up to 2 years post-intervention
Population: All patients were MRD negative at the end of Induction I. No patients were assigned low risk due to low risk molecular and cytogenetic features. All high risk patients had high risk molecular and cytogenetic features.
Measure: Median (Full Range); unit: years
Groups:
- Patients Who Are MRD Negative: Patients who are MRD negative but lack high or low risk molecular and cytogenetic features, defined as time from end of first course of therapy to death or relapse.
Arm/Group | Patients Who Are MRD Negative
Number analyzed (Participants) | 5
years | 1.08 [0.04 to NA] — Insufficient number of participants with events; maximum observation was censored at last follow-up.

5. Secondary Outcome: Cardiotoxicity in Patients With de Novo AML That Receive the Four-cycle Aflac-AML Regimen With the Inclusion of Dexrazoxane
Description: Number of patients that develop cardiac ejection fraction <50% (CTCAE V5.0 grade 2 or greater dysfunction) either during therapy (early cardiotoxicity) or after completion of therapy (late cardiotoxicity)
Time Frame: At completion of Cycle 4 (each cycle average is 28 days)
Population: The definition of late cardiotoxicity is after completion of therapy. All 3 of the high risk patients came off protocol early and did not complete therapy. For the low risk patients, 2 did not complete therapy. Among the 3 that did complete therapy, 1 patient has been lost to follow-up since completion of therapy with no cardiac data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflac-AML Low Risk Patients | Aflac-AML High Risk Patients
Number analyzed (Participants) | 5 | 3
Participants
  Early cardiotoxicity | 0 | 0
  Late cardiotoxicity: number analyzed (Participants) | 2 | 0
  Late cardiotoxicity | 0 | 0

6. Secondary Outcome: Proportion of Patients Who Develop Infection and/or Febrile Neutropenia During Each Treatment Course
Description: Number of participants that developed infection and/or febrile neutropenia at the end of each treatment cycle.
Time Frame: At the end of each cycle (each cycle average is 28 days)
Population: All 3 of the high risk patients came off protocol early and did not complete therapy. For the low risk patients, 2 did not complete therapy. Among the 3 that did complete therapy, 1 patient has been lost to follow-up since completion of therapy with no cardiac data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflac-AML Low Risk Patients | Aflac-AML High Risk Patients
Number analyzed (Participants) | 5 | 3
Participants
  Cycle 1 - Induction 1 | 5 | 2
  Cycle 2 - Induction 2 | 3 | 2
  Cycle 3 - Induction 3: number analyzed (Participants) | 3 | 0
  Cycle 3 - Induction 3 | 2 | 0
  Cycle 4 - Induction 4: number analyzed (Participants) | 3 | 0
  Cycle 4 - Induction 4 | 2 | 0

7. Secondary Outcome: Duration of Hospital Admission in Patients That Developed Infection and Febrile Neutropenia at the End of Each Treatment Cycle
Description: Duration of hospital admission in patients that developed infection and febrile neutropenia at the end of each treatment cycle
Time Frame: At the end of each cycle (each cycle average is 28 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Aflac-AML Low Risk Patients | Aflac-AML High Risk Patients
Number analyzed (Participants) | 5 | 2
days
  Cycle 1 - Induction 1 | 33 (5.1) | 30 (5.7)
  Cycle 2 - Induction 2: number analyzed (Participants) | 3 | 2
  Cycle 2 - Induction 2 | 29.3 (1.5) | 30.0 (1.4)
  Cycle 3 - Induction 3: number analyzed (Participants) | 2 | 0
  Cycle 3 - Induction 3 | 29 (5.7) |
  Cycle 4 - Induction 4: number analyzed (Participants) | 2 | 0
  Cycle 4 - Induction 4 | 27.5 (0.7) |

ADVERSE EVENTS:
Time Frame: Time of consent through end of follow-up (Up to 2 years post-intervention).
Groups:
- Induction I: Participants in this group received AraC/Daunorubicin/Etoposide (10+3+5) +/- GO based on CC genotype^ Patients were classified into risk groups following Induction I
  * ^If has FLT3-ITD mutation, Sorafenib is added
- Low Risk - Induction II: Participants in this group received Mitoxantrone/AraC
- High Risk - Induction II: Participants in this group received Mitoxantrone/AraC^
  * ^If has FLT3-ITD mutation, Sorafenib is added
- Low Risk - Intensification I: Participants in this group received AraC/Etoposide
- Low Risk - Intensification II: Participants in this group received HD AraC/Asparaginase
Arm/Group | Induction I | Low Risk - Induction II | High Risk - Induction II | Low Risk - Intensification I | Low Risk - Intensification II
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 8/8 | 5/5 | 3/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction I (N=8) | Low Risk - Induction II (N=5) | High Risk - Induction II (N=3) | Low Risk - Intensification I (N=3) | Low Risk - Intensification II (N=3)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 8 (8) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Lymphocyte Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Platelet count decreased (Investigations) | 6 (6) | 4 (4) | 2 (2) | 3 (3) | 3 (3)
White Blood Cell Decreased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Weight loss (Investigations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04326439/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT04326439/ICF_001.pdf